CLINICAL TRIAL: NCT04329858
Title: the Antibacterial Effect of Different Glass Ionomer Restoration Containing Zinc ,Silver and Fluoride Ion:in Situ Study
Brief Title: the Antibacterial Effect of Zinc ,Silver and Fluoride
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina mounir elkady, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6679
Record Dates: First submitted 2018-07-17; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- conventional glass ionomer (Active Comparator)
  Interventions: Procedure: conventional glass ionomer
- zinc modified glass ionomer (Experimental)
  Interventions: Procedure: zinc modified
- silver modified glass ionomer (Experimental)
  Interventions: Procedure: silver modified glass ionomer

INTERVENTIONS:
Procedure: silver modified glass ionomer — occlusal cavity filled with silver modified
  Arms: silver modified glass ionomer
Procedure: zinc modified — occlusal cavity filled with zinc modified
  Arms: zinc modified glass ionomer
Procedure: conventional glass ionomer — occlusal cavity filled with conventional glass ionomer
  Arms: conventional glass ionomer

SUMMARY:
natural teeth will be filled with the 3 different material then the dentin sample will be collected ,bacterial culture and elementary analysis will be done

DETAILED DESCRIPTION:
orthodontic patient with premolar indicated for extraction , teeth will restored with the different material 3 months before doing extraction

ELIGIBILITY:
Inclusion Criteria:

* patient need teeth extraction for orthodontic treatment

Exclusion Criteria:

* carious teeth deciduous teeth

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
bacterial count | 3months
  streptococcus mutant count by culture of dentin sample excavated from the tooth after restoration removal
elementary analysis of dentin | 3months
  elementary analysis of dentin component excavated from the cavity after restoration removal to detect the change in tooth mineral